CLINICAL TRIAL: NCT06827873
Title: Effect of Oral Supplement Intervention on Influenza Vaccine Efficacy: a Randomized Controlled Clinical Trial
Brief Title: Effect of Oral Supplements for Influenza Vaccine Response
Acronym: EOSIIVE-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tsinghua University (Other)
Collaborators: Second Affiliated Hospital of Bengbu Medical College (Other)
Responsible Party: Principal Investigator, Ai Zhao, Associate Professor, Tsinghua University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: THU01-20240201
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Influenza Vaccine Response
Keywords: Vaccine Efficacy; Elderly Immunity; Fatty Acid Supplementation; Gut Microbiota; Randomized Controlled Trial
MeSH Terms: interventions — Arachidonic Acid; Dietary Supplements; ursodoxicoltaurine; Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Forty-five adults aged 60-70 years are randomly assigned in equal numbers (n=15 per group) to three parallel groups: two intervention groups receiving different supplements(arachidonic acid and TUDCA) and one control group receiving placebo. The intervention period lasts 25 days, from Day 0 to Day 24. Triple-blinding is implemented to ensure that both participants and investigators are unaware of group assignments.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study supplements are identical in appearance and packaging to maintain blinding.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ARA (Arachidonic Acid) Supplement Group (Experimental): Participants will take 1000 mg of ARA (Arachidonic Acid) dietary supplement capsules daily. Maintain original lifestyle during intervention, Day 0-Day 2 as adaptation period, receive quadrivalent influenza vaccine on Day 3, continue supplementation until Day 24.
  Interventions: Dietary Supplement: ARA (Arachidonic Acid) Supplementation; Biological: Shanghai Biological Quadrivalent Influenza Virus Inactivated Vaccine
- TUDCA (Tauroursodeoxycholic acid) Supplement Group (Experimental): Participants will take 1000 mg of TUDCA (Tauroursodeoxycholic acid) dietary supplement capsules daily. Capsules primarily contain TUDCA, with 500 mg per serving (two capsules). Maintain original lifestyle during intervention, Day 0-Day 2 as adaptation period, receive quadrivalent influenza vaccine on Day 3, continue supplementation until Day 24.
  Interventions: Drug: TUDCA (Tauroursodeoxycholic Acid) Supplementation; Biological: Shanghai Biological Quadrivalent Influenza Virus Inactivated Vaccine
- Placebo Comparator Group (Placebo Comparator): Participants will take 1000 mg of placebo capsules identical in appearance and smell. Maintain original lifestyle during intervention, Day 0-Day 2 as adaptation period, receive quadrivalent influenza vaccine on Day 3, continue taking placebo until Day 24.
  Interventions: Dietary Supplement: Placebo Supplementation; Biological: Shanghai Biological Quadrivalent Influenza Virus Inactivated Vaccine

INTERVENTIONS:
Dietary Supplement: ARA (Arachidonic Acid) Supplementation — Oral ARA (Arachidonic Acid) dietary supplement capsules, dosage 1000 mg/person/day. Capsule composition includes: C14:0 (0.15%), C16:0 (6.08%), C16:1 (0.15%), C18:0 (4.57%), C18:1 (19.65%), C18:2 (38.46%), C18:3 (0.87%), C20:0 (0.50%), C20:3 (2.00%), C20:4 (18.66%), C22:0 (1.81%), C24:0 (4.05%). Maintain original lifestyle during intervention, Day 0-Day 2 as adaptation period, receive quadrivalent influenza vaccine on Day 3, continue supplementation until Day 24.
  Other Names: AA; 5,8,11,14-Eicosatetraenoic acid; C20:4
  Arms: ARA (Arachidonic Acid) Supplement Group
Drug: TUDCA (Tauroursodeoxycholic Acid) Supplementation — Oral Double Wood brand TUDCA (Tauroursodeoxycholic Acid) dietary supplement capsules, dosage 1000 mg/person/day. Capsules primarily contain TUDCA, with 500 mg per serving (two capsules), other ingredients include gelatin and rice powder. Maintain original lifestyle during intervention, Day 0-Day 2 as adaptation period, receive quadrivalent influenza vaccine on Day 3, continue supplementation until Day 24.
  Arms: TUDCA (Tauroursodeoxycholic acid) Supplement Group
Dietary Supplement: Placebo Supplementation — Oral placebo capsules identical in appearance and smell, dosage 1000 mg/person/day. Placebo capsule composition includes: C14:0 (0.09%), C16:0 (6.12%), C16:1 (0.03%), C18:0 (3.50%), C18:1 (28.06%), C18:2 (59.40%), C20:0 (0.27%), C22:0 (0.76%), C24:0 (0.26%). Maintain original lifestyle during intervention, Day 0-Day 2 as adaptation period, receive quadrivalent influenza vaccine on Day 3, continue taking placebo until Day 24.
  Other Names: Placebo Capsules
  Arms: Placebo Comparator Group
Biological: Shanghai Biological Quadrivalent Influenza Virus Inactivated Vaccine — Administer Shanghai Biological Quadrivalent Influenza Virus Inactivated Vaccine, produced by Shanghai Biological Products Research Institute Co., Ltd. , specification 0.5ml/dose, containing 15.0 μg hemagglutinin (for each influenza virus strain), suitable for intramuscular injection in individuals 6 months and older. Administer one dose to all study participants on Day 3. Closely observe and record any potential adverse reactions after vaccination.
  Other Names: Quadrivalent Influenza Vaccine

SUMMARY:
The aim of this clinical trial is to explore the efficacy of fatty acid and bile acid based supplements on enhancing influenza vaccine immune response in adults aged 60-70 years. The objectives of this study are:

1. To explore the efficacy of fatty acid and bile acid based supplements on enhancing flu vaccine immune response.
2. To evaluate the safety of fatty acid and bile acid use in elders.
3. To explore the potential role of microbiota in regulating immune response.

This study will conduct a randomized clinical trial to compare the efficacy of fatty acid / bile acid (Tauro Ursodesoxy Cholic Acid, TUDCA)supplements on enhancing vaccine immune response. The antibody's titer and safety indicators after influenza vaccination will be evaluated. Study process are:

1. Participants will be required to intake the assigned supplement or placebo daily for 25 days;
2. Receive a influenza vaccine on day 4;
3. Provide blood samples three times and stool samples twice at base line and endpoint respectively;
4. The antibody's titer and safety indicators will be analyzed and compared among groups.

This study aims to establish a theoretical foundation for utilizing nutritional strategies to enhance vaccine-induced immune responses and to provide a scientific framework for developing oral vaccine boosters.

DETAILED DESCRIPTION:
Influenza virus infection presents a significant global health challenge, particularly threatening the elderly population due to immunosenescence. The immune response to influenza vaccination involves a complex series of events: after vaccination, hemagglutination inhibition antibody titers peak around day 14, accompanied by the production of neutralizing antibodies and other specific antibodies. This immune response gradually stabilizes to a post-response baseline level as immune memory establishes.

The age-related decline in immune function manifests through multiple mechanisms,including: reduced production of naive T cells; decreased diversity of T cell repertoire; compromised B cell function, altered cytokine production profiles which all diminished vaccine response efficacy.

Recent advances in immunometabolism have revealed the crucial role of specific fatty acids in immune system modulation. Our preliminary explorations found that，short-term Arachidonic Acid（AA）intervention could significantly reduce the time required for antibody production and enhance its levels following rabies vaccination. We also noticed that the serum Tauro Ursodesoxy Cholic Acid (TUDCA) was elevated in the intervention group. However, the related mechanism is still not clear.

The theoretical framework integrates nutritional immunology with classical vaccinology, focusing on the metabolic interaction between dietary fatty acids and immune cell function. This approach is particularly relevant for the elderly population, where reduced vaccine responsiveness due to immunosenescence presents a significant challenge in achieving optimal vaccine protection.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60-70 years old
2. Body Mass Index (BMI) 18.5-26.9 kg/m²
3. No influenza vaccination in the past year
4. Able to understand and sign the informed consent form, and capable of completing the full follow-up process

Exclusion Criteria:

1. Severe lipid metabolism disorders
2. Use of lipid-lowering medications, weight loss drugs, or insulin within the past three months
3. Vaccination with other vaccines within the past three months
4. Use of probiotics or prebiotics within the past three months
5. Use of steroids, immunosuppressants, or other hormonal medications within the past year
6. Immunodeficiency diseases
7. Severe vaccine allergy history
8. Liver or kidney metabolic disorders
9. Occurrence of fever, common cold, severe diarrhea, or other diseases within the past month
10. Poorly controlled chronic diseases (such as blood pressure, blood sugar)
11. Intake of influenza antiviral drugs within the past two weeks
12. Cognitive function impairment
13. Planning to undergo surgery in the near future

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Specific Antibody Levels and Neutralizing Antibody Responses to Influenza Vaccine | Day 13 and Day 24
  By detecting serum neutralizing and specific antibody levels on Day 13 and Day 24, evaluate the impact of different dietary supplements on influenza vaccine immune responses in elderly individuals. Focus primarily on changes in antibody titers to determine whether dietary supplementation can enhance vaccine immunogenicity.

SECONDARY OUTCOMES:
Changes in Inflammatory Markers | Day 0 and Day 24
  Measure serum levels of inflammatory factors such as IL-1, IL-2, IL-6, IL-8, IL-10, IL-17 to assess the potential modulatory effect of dietary supplementation on inflammatory responses.
Gut Microbiota Composition Changes | Day 0 and Day 24
  Analyze intestinal microbiota structure and metabolomics changes through fecal samples to explore the impact of dietary supplementation on gut microecology, including:
  1. Alpha diversity analysis (Shannon index, Chao1 index, observed species)
  2. Beta diversity analysis (UniFrac distance, Bray-Curtis dissimilarity)
  3. Microbial species composition and relative abundance changes
  4. Key microbiota (such as Bacteroidetes, Actinobacteria) abundance analysis
  5. Metabolic pathway changes, including KEGG functional pathway prediction and microbiota-related immune metabolic pathways
Metabolomics Analysis | Day 0, Day 13 and Day 24
  Perform non-targeted metabolomics detection to evaluate the impact of dietary supplementation on human metabolic levels, including lipid profiles, liver and kidney function indicators.

OTHER OUTCOMES:
Safety Assessment | Throughout the entire study period (Day 0-Day 24)
  Record and analyze adverse reactions during the intervention, including clinical symptoms, blood routine, and biochemical indicators to assess the safety of dietary supplements.
Dietary Intake Assessment | Day 0 and Day 24
  Record dietary intake patterns of study subjects through 24-hour dietary recall and FFQ surveys to control nutritional factors that might influence results.
Coagulation Function and Thrombosis Risk Assessment | Day 0 and Day 24
  Assess the impact of dietary supplements on blood coagulation function by detecting coagulation time and related coagulation indicators, and exclude the risks of coagulation disorders and thrombosis. Focus on changes in coagulation time, platelet count, and coagulation factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Tsinghua University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sainz T, Casas I, Gonzalez-Esguevillas M, Escosa-Garcia L, Munoz-Fernandez MA, Prieto L, Gosalbes MJ, Jimenez-Hernandez N, Ramos JT, Navarro ML, Mellado MJ, Serrano-Villar S, Calvo C. Nutritional Supplementation to Increase Influenza Vaccine Response in Children Living With HIV: A Pilot Clinical Trial. Front Pediatr. 2022 Jul 19;10:919753. doi: 10.3389/fped.2022.919753. eCollection 2022. PMID 35928688
- [Result] D'Onofrio V, Porrez S, Jacobs B, Alhatemi A, De Boever F, Waerlop G, Michels E, Vanni F, Manenti A, Leroux-Roels G, Platenburg PP, Hilgers L, Leroux-Roels I. Safety and Immunogenicity of a Carbohydrate Fatty Acid Monosulphate Ester Adjuvant Combined with a Low-Dose Quadrivalent Split-Virion Inactivated Influenza Vaccine: A Randomised, Observer-Blind, Active-Controlled, First-in-Human, Phase 1 Study. Vaccines (Basel). 2024 Sep 10;12(9):1036. doi: 10.3390/vaccines12091036. PMID 39340066
- [Result] Chou CH, Mohanty S, Kang HA, Kong L, Avila-Pacheco J, Joshi SR, Ueda I, Devine L, Raddassi K, Pierce K, Jeanfavre S, Bullock K, Meng H, Clish C, Santori FR, Shaw AC, Xavier RJ. Metabolomic and transcriptomic signatures of influenza vaccine response in healthy young and older adults. Aging Cell. 2022 Sep;21(9):e13682. doi: 10.1111/acel.13682. Epub 2022 Aug 23. PMID 35996998

DOCUMENTS (1):
  • Informed Consent Form (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT06827873/ICF_000.pdf